CLINICAL TRIAL: NCT04612712
Title: A Phase 1/2 Dose Escalation and Expansion Study of Donafenib Tosilate Tablets in Combination With KN046 Injection in Advanced Gastrointestinal Tumors
Brief Title: A Phase 1/2 Study of Donafenib in Combination With KN046 in Advanced Gastrointestinal Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Collaborators: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN046D-C-101
Record Dates: First submitted 2020-10-29; First posted 2020-11-03 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Advanced Gastrointestinal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib+ KN046 (Experimental): Donafenib 50mg BID/100 mg BID/200 mg BID orally + KN046 5mg/kg Q3W iv
  Interventions: Drug: Donafenib Tosilate Tablets; Biological: KN046 Injection

INTERVENTIONS:
Drug: Donafenib Tosilate Tablets — In the dose exploration phase (phase I) : three doses of Donafenib tosylate tablets [50 mg twice a day; 100 mg twice a day; 200 mg twice a day ] will be explored. In the dose expansion phase (phase II), patients with advanced hepatocellular carcinoma will be treated at the recommended dose for phase 2(RP2D).The RP2D will be determined by the dose escalation study.
Biological: KN046 Injection — 5mg/kg Q3W

SUMMARY:
This study is an open, multi-center clinical trial, the purpose is to study the safety and preliminary efficacy of Donafenib combined with KN046 in subjects with Advanced Gastrointestinal Tumors.

DETAILED DESCRIPTION:
The study consists of dose escalation and dose expansion. The preset dose of Donafenib is 50 mg BID, 100 mg BID and 200 mg BID, and the preset dose of KN046 is 5 mg/kg Q3W. Dose expansion will enroll subjects who with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-70 years;
* Phase I dose escalation: Advanced gastric cancer, esophageal cancer, colorectal cancer, hepatocellular carcinoma, pancreatic cancer (other than pancreatic neuroendocrine tumors) and intrahepatic cholangiocarcinoma that failed standard treatments confirmed by histopathology and/or cytology; Among them, the Child-Pugh score of liver function in patients with hepatocellular carcinoma is less than 5,
* Phase II advanced hepatocellular carcinoma Dose expansion: Patients with advanced hepatocellular carcinoma who are clinically diagnosed or confirmed by histopathology and/or cytology and are not suitable for surgical resection; The patient has not undergone first-line systemic treatment [small molecule targeted drugs (such as sorafenib, lenvatinib, etc.), systemic chemotherapy] and tumor immunotherapy (anti-PD-1/L1, CTLA-4, etc.); Child-Pugh score of liver function ≤ 6;
* Has at least one measurable lesion based on RECIST 1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* Life expectancy ≥12 weeks;
* Patients must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Subjects who have previously received immune checkpoint inhibitors (such as anti-PD-1/L1, CTLA-4, etc.);
* History of interstitial lung disease or non-infectious pneumonia;
* Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or patients undergoing total gastrectomy;
* Has received vaccination within 4 weeks prior to the first dose.
* Has participated in other anticancer drug clinical trials within 4 weeks.
* According to the judgement of the investigators, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Phase I part - Tolerability of Donafenib in Combination With KN046 | 21 days after the first dose of Donafenib and KN046
  Evaluated by severity of drug-related adverse events (AEs), serious adverse events (SAEs).
Phase II part - Objective response rate(ORR) | From the time of initial administration until intolerant toxicity, disease progression, withdrawal of ICF, loss of follow-up, death or early study termination occurs (whichever occurs first),assessed up to 36 months]
  Objective response rate based on the RECIST 1.1 by investigator. Percentage of subjects achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Duration of Response (DOR) | Through study completion, an expected average of 3 year
  It is defined as time between the date of first radiographic documented objective response and the date of the radiographic documented disease progression.
Progression-Free Survival (PFS) | Through study completion, an expected average of 3 year
  PFS is defined as the time from date of enrollment to the date of the first objectively documented tumor progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, PhD, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No